CLINICAL TRIAL: NCT04007016
Title: A New Pelvic Osteotomy Method for Open Reduction in the Treatment of Developmental Dysplasia of the Hip in Children
Brief Title: A New Pelvic Osteotomy Method for Open Reduction
Status: Completed | Type: Observational
Sponsor: Yuxi Su (Other)
Responsible Party: Sponsor-Investigator, Yuxi Su, Vice Professor of Pediatric orthopedic, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: Yuxi-Guoxin 201906
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pemberton osteotomy （PO）: PO group received Pemberton osteotomy
- inner "L shaped" iliac osteotomy (ILSO): ILSO group received inner "L shaped" iliac osteotomy
  Interventions: Procedure: a new osteotomy from the inner "L shaped" iliac osteotomy

INTERVENTIONS:
Procedure: a new osteotomy from the inner "L shaped" iliac osteotomy — There were two ostectomies were used in the osteotomy. The first was was a cured and 5mm width and the second one was straight 1.5cm width. All the directions was started from the inner to outer just a bove the triradiate cartilage and its shape like"L"
  Groups: inner "L shaped" iliac osteotomy (ILSO)

SUMMARY:
Developmental dysplasia of the hip (DDH) was one of the most common hip disorders disease in children. Pemberton osteotomy (PO) was one of the most widely used by the pediatric orthopedic surgeons. In our clinical work, the investigators found some defect the operation procedure. When the surgeons were not familiar to the PO, it may injured the triradiate cartilage or easily be absorbable of the distal iliac. Here, the investigators found a new pelvic osteotomy just from the inner "L shaped" iliac osteotomy (ILSO) to treat DDH. This approach was in a visible part of the sciatic notch and not presumed to be in the ischium, completely out of sight. Comparing to the PO method, the investigators' operation method was easy to master and had less complications.

ELIGIBILITY:
Inclusion Criteria:

* over two years old
* open reduction and acetabular osteotomy
* diagnosed as developmental dysplasia of the hip

Exclusion Criteria:

* a previous history of DDH surgery
* teratologic dislocations
* cerebral palsy
* other spastic or neuromuscular disease

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients were evaluated and treated in the same hospital and the same surgeon did all the operation. The study was carried out between Mar 2016 and May 2018.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
preoperative acetabular index | 6th month after surgery
  preoperative acetabular index by measure the postoperative X-ray
Wiberg's mean center-edge angle | 6th month after surgery
  center-edge angle by measure the postoperative X-ray

SECONDARY OUTCOMES:
blood loss | 1st day after surgery
  blood loss during surgery
avascular necrosis (AVN) | through study completion, an average of 1 year
  avascular necrosis (AVN) of the femoral head according to the Kalamchi and McEwen classification

IPD SHARING:
Plan to Share IPD: Undecided